CLINICAL TRIAL: NCT00052429
Title: Phase I/II Study of Dose-Painting Using Intensity Modulated Radiation Therapy Plus Chemotherapy in Patients With Stage II-IVB Nasopharyngeal Carcinoma
Brief Title: High-Dose Radiation Therapy Plus Chemotherapy in Treating Patients With Advanced Nose or Throat Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-077; MSKCC-02077; NCI-H02-0101
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Head and Neck Cancer
Keywords: stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Fluorouracil; Chemotherapy, Adjuvant; Radiotherapy

ARMS (1):
- High-Dose Radiation Therapy Plus Chemotherapy (Experimental): Phase I
  * Radiotherapy: Patients receive radiotherapy once daily 5 days a week for 6 weeks beginning on day 1.
  * Concurrent chemotherapy: Patients receive cisplatin IV over 20-30 minutes on days 1-5 and 22-26.
  * Adjuvant chemotherapy: Approximately 2-5 weeks after the completion of radiotherapy, patients receive fluorouracil IV continuously on days 1-4 and cisplatin IV over 20-30 minutes on days 1-5 and 22-26. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. In the absence of dose-limiting toxicity in 1 whole cohort of patients, study proceeds to phase II. Phase II
  * Patients are treated as in phase I. Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.
  Interventions: Drug: cisplatin; Drug: fluorouracil; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining high-dose radiation with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining high-dose radiation therapy with chemotherapy in treating patients who have newly diagnosed stage II, stage III, or stage IV nasopharyngeal cancer.

DETAILED DESCRIPTION:
OUTLINE: Cohorts of 10 patients receive the following treatment to assess for dose-limiting toxicity.

Phase I

* Radiotherapy: Patients receive radiotherapy once daily 5 days a week for 6 weeks beginning on day 1.
* Concurrent chemotherapy: Patients receive cisplatin IV over 20-30 minutes on days 1-5 and 22-26.
* Adjuvant chemotherapy: Approximately 2-5 weeks after the completion of radiotherapy, patients receive fluorouracil IV continuously on days 1-4 and cisplatin IV over 20-30 minutes on days 1-5 and 22-26. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

In the absence of dose-limiting toxicity in 1 whole cohort of patients, study proceeds to phase II.

Phase II

* Patients are treated as in phase I. Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nasopharyngeal cancer

  * Stage II-IVB
  * Newly diagnosed
* No distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* AST no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Calcium no greater than 11.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Medically able to tolerate a definitive course of radiotherapy and the necessary immobilization
* No other active malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for this diagnosis
* More than 3 years since other prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for this diagnosis
* More than 3 years since other prior radiotherapy
* No prior radiotherapy to the head and neck region

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Wolden, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Bakst RL, Lee N, Pfister DG, Zelefsky MJ, Hunt MA, Kraus DH, Wolden SL. Hypofractionated dose-painting intensity modulated radiation therapy with chemotherapy for nasopharyngeal carcinoma: a prospective trial. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):148-53. doi: 10.1016/j.ijrobp.2010.01.026. Epub 2010 Jun 3. PMID 20605352
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Dose Radiation Therapy Plus Chemotherapy
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High-Dose Radiation Therapy Plus Chemotherapy
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate of Patients
Description: Patients will be followed indefinitely and will have standard screening for development of distant metastases, including physical exam, as well as liver function tests and a chest radiograph annually. Patients will be classified as progression free as long as they remain alive with local, regional or distant recurrence.
Time Frame: up to 77 months
Measure: Median (Full Range); unit: months
Arm/Group | High-Dose Radiation Therapy Plus Chemotherapy
Number analyzed (Participants) | 25
months | 33 [14 to 77]

2. Primary Outcome: Local Control of Participants
Description: Patients will be classified as controlled as long as there is no clinical or radiographic evidence of disease progression. Physical exam with fiberoptic nasopharyngoscopy will be performed approximately every 3 months in the first year of follow-up, every 4 months in the second year, every 6 months in the third-fifth years and annually, thereafter.
Time Frame: every 3 months in the first year of follow-up, every 4 months in the second year, every 6 months in the third-fifth years and annually, thereafter.
Measure: Number; unit: percentage of participants
Arm/Group | High-Dose Radiation Therapy Plus Chemotherapy
Number analyzed (Participants) | 25
percentage of participants
  Actuarial rate of local control | 91
  Regional control | 91
  Metastases-free survival | 91
  Overall survival | 89

ADVERSE EVENTS:
Arm/Group | High-Dose Radiation Therapy Plus Chemotherapy
Serious Adverse Events (participants affected / at risk) | 19/25
Other Adverse Events (participants affected / at risk) | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Radiation Therapy Plus Chemotherapy (N=25)
Central nervous system necrosis (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4)
Fever (General disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (4)
Infectious meningitis (Infections and infestations) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Mucositis-Oral cavity (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decrease (Investigations) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Chills (General disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Syncope (Nervous system disorders) | 2 (2)
Renal and urinary disorders -Other, specify-Renal tubular disorder (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Radiation Therapy Plus Chemotherapy (N=25)
Ear disorder (Ear and labyrinth disorders) | 2 (2)
Fatigue (General disorders) | 4 (6)
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Mucositis-Oral (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes